CLINICAL TRIAL: NCT01994200
Title: Developing and Implementing an Interdisciplinary Team-Based Care Approach (ITCA-ThyCa) For Newly Diagnosed Thyroid Cancer Patients: Randomized Controlled Trial
Brief Title: Developing and Implementing an Interdisciplinary Team-Based Care Approach (ITCA-ThyCa) for Thyroid Cancer Patients
Acronym: ITCA-ThyCa
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Melissa Henry, Assistant Professor and Psychologist, Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GZ-2013-10963
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Thyroid Cancer
Keywords: Thyroid cancer; New diagnosis; Dedicated Nurse; Interdisciplinary team; Randomized Controlled Trial; Intervention; Supportive care
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interdisciplinary Team-Based Approach (Experimental): The delivered intervention will be to provide patients with an interdisciplinary team-based approach defined as care provided by a variety of professionals, each having their own domain of expertise, defined roles and responsibilities, who work together and meet to discuss patient needs and develop comprehensive treatment plans. Team composition will include physicians, a dedicated nurse, and allied professionals (e.g., dieticians, social workers, psychologists). The dedicated nurse will have a central integrative role in this interdisciplinary team and will provide patients with information about their illness and treatment, symptom management, emotional support, and reference to other resources when needed
  Interventions: Other: Interdisciplinary Team-Based Approach
- Usual Care Control Group (Other): Patients in the control group will be provided with usual care, comprised of meetings with surgeons and endocrinologists. All patients in this study will be provided with an information website containing information on their cancer, treatments, and treatment side-effects.
  Interventions: Other: Usual Care Control

INTERVENTIONS:
Other: Interdisciplinary Team-Based Approach — Three meetings will be scheduled with the oncology dedicated-nurse. First meeting: information about the physical illness; the emotional impact of being newly diagnosed with thyroid cancer; as well as surgery and its' short- and long-term consequences. Second meeting: information on radioactive iodine treatments and its associated safety precautions, nutrition and dietary considerations. Third meeting: how the cancer diagnosis can be an opportunity to make important lifestyle changes and establish new life-priorities. The dedicated nurse, in collaboration with the Department of Nursing and ENT, will develop and implement an interdisciplinary team-based approached developed for this study according to guidelines of the Programme québécois de lutte contre le cancer (PQLC).
  Other Names: Interdisciplinary Team-Based Approach (ITCA-ThyCa)
  Arms: Interdisciplinary Team-Based Approach
Other: Usual Care Control — Patients in the control group will be provided with usual care, comprised of meetings with surgeons and endocrinologists. All patients in this study will be provided with an information website containing information on their cancer, treatments, and treatment side-effects.
  Arms: Usual Care Control Group

SUMMARY:
While thyroid cancer is generally associated with a favourable prognosis, there is a discrepancy with how important if not traumatic its impact can be on patients. Quality of life (QoL) decreases in the year following a thyroid cancer diagnosis, constituting an optimal period for a preventive intervention. The goal of this study is to evaluate the impact of offering an interdisciplinary team-based care approach for newly diagnosed thyroid cancer patients, including a dedicated nurse who will provide important psychoeducational elements identified in previous focus group studies of thyroid cancer patients, i.e., information on: the physical illness; the emotional impact of being newly diagnosed with thyroid cancer; surgery and its' short- and long-term consequences; radioactive iodine treatments and its associated safety precautions, nutrition and dietary considerations; and how the cancer diagnosis can be an opportunity to make important lifestyle changes and establish new life-priorities.

DETAILED DESCRIPTION:
The investigators will conduct a 2-arm Randomized Controlled Trial comparing an Interdisciplinary Team-Based Care Approach to usual care.

The primary research question will be: Does adding the Interdisciplinary Team-Based Care Approach (ITCA-ThyCa) to usual care (EG) increase levels of overall QoL among newly diagnosed thyroid cancer patients, compared with those receiving usual care (UC), at 9 months post-randomization (i.e., after all of the dedicated-nurse meetings are administered) as judged by scores on the Functional Assessment of Chronic Illness Therapy-General (FACT-G)? Primary hypothesis: The EG will report higher scores of overall QoL on the FACT-G than the UC at 9 months post-randomization.

Secondary research questions: The investigators plan to evaluate ITCA-ThyCa effects on secondary outcomes such as level of: physical health (SF-36 Physical Health subscale), mental health (SF-36 Mental Health subscale), fatigue (Functional Assessment of Chronic Illness Therapy-Fatigue; FACIT-F), anxiety and depression (Hospital Anxiety and Depression Scale; HADS), and negative illness perception (Illness Perception Questionnaire - Revised (IPQ-R). The investigators also plan to explore ITCA-ThyCa effects on satisfaction with care (16 questions of the NRC Picker satisfaction survey measuring patient satisfaction with care) and healthcare service use (types of professionals consulted, frequency of visits, and time elapsed between referral and first consultation). Hypotheses: The EG will report a higher level of physical and mental health on the SF-Physical and Mental Health subscales, respectively; and a lower level of fatigue on the FACIT-F, anxiety and depression on the HADS, and negative illness perception on the IPQ-R; compared with the UC at 9 months post-randomization.

All of the abovementioned changes will be present throughout the treatment, namely at 7-10 days and 5 months post-randomization (i.e., immediately after each of the meetings planned with the dedicated nurse).

All of the abovementioned changes will persist at 12 months post-randomization (i.e., corresponding to 6 months after all anti-cancer treatments are completed and 3 months after all dedicated-nurse meetings have been administered).

Feasibility and acceptability (9 first months of the trial):

The investigators plan on testing the feasibility and acceptability of the 2-arm RCT of ITCA-ThyCa during the first 9 months of the trial (once the investigators start recruiting, after the first 3-6 months dedicated to hiring our personnel and developing the manual of our approach). During this phase, the investigators will aim to address the following research questions:

1. Can the investigators recruit a sufficient number of patients (i.e., a minimum of 60 patients over 6 months or 10/month) and retain a sufficient proportion of thyroid cancer patients (i.e., at least 80% at 7-10 days, 5 months or 9 months post-randomization) in both trial arms?
2. Is ITCA-ThyCa acceptable to at least 80% of EG thyroid cancer patients? Secondary pilot study questions
3. Which evaluation time should be primary post-randomization, based on an acceptable retention rate of 80%?
4. What variance estimates can be used to inform calculation of sample size for the full study?

If the design remains the same following this pilot, the investigators aim to roll in the pilot data in the full trial.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with a first occurrence of thyroid cancer <2-4 weeks of diagnosis (i.e., histologically confirmed thyroid cancer (papillary, follicular, or medullary type; TNM classification system);
* Willing to participate in the EG meetings;
* >18 years;
* Alert and capable of giving free and informed consent;
* Able to speak and read English or French.

Exclusion Criteria:

* Anaplastic thyroid cancer;
* Karnofsky Performance Status (KPS) score <60 (rated by the Research Coordinator (RC) or referring physician) or expected survival <6 months according to clinical judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Overall quality of life | 9 months post-randomization
  Measure: Functional Assessment of Chronic Illness Therapy-General (FACT-G)

SECONDARY OUTCOMES:
Level of physical health | 9 months post-randomization
  Measure: SF-36 Physical Health subscale
Level of mental health | 9 month post-randomization
  Measure: SF-36 Mental Health subscale
Level of fatigue | 9 months post-randomization
  Measure: Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F)
Level of anxiety and depression (combined) | 9 month post-randomization
  Measure: Hospital Anxiety and Depression Scale (HADS)
Level of negative illness perception | 9 month post-randomization
  Illness Perception Questionnaire - Revised (IPQ-R)
Level of satisfaction with care | 9 month post-randomization
  16 questions of the NRC Picker satisfaction survey measuring patient satisfaction with care
Healthcare service use | Over 9 months post-randomization
  Types of professionals consulted, frequency of visits, and time elapsed between referral and first consultation

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Henry, PhD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada